CLINICAL TRIAL: NCT05519046
Title: Clinical and Functional Effects of Cardiac Contractility Modulation in Chagas Heart Disease: a Randomized Study - Contractility - FIX-Chagas
Brief Title: Cardiac Contractility Modulation in Chagas Heart Disease
Acronym: FIX-Chagas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Collaborators: Impulse Dynamics (Industry); I2medi Comercial Medica LTDA (Unknown)
Responsible Party: Principal Investigator, Martino Martinelli Filho, Principal Investigator, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 57563722.3.0000.0068
Record Dates: First submitted 2022-08-10; First posted 2022-08-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chagas Cardiomyopathy; Heart Failure; Systolic Dysfunction; Right Bundle Branch Block and Left Anterior Fascicular Block; Right Bundle Branch Block and Left Posterior Fascicular Block
MeSH Terms: conditions — Chagas Cardiomyopathy; Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac Contractility Modulation Group - CCM Group (Experimental): CCM implantation.
  Interventions: Device: Cardiac Contractility Modulation (CCM)
- Cardiac Resynchronization Therapy Group - CRT Group (Active Comparator): CRT implantation
  Interventions: Device: CRT

INTERVENTIONS:
Device: Cardiac Contractility Modulation (CCM) — Cardiac Contractility Modulation (CCM) implantation
  Arms: Cardiac Contractility Modulation Group - CCM Group
Device: CRT — Cardiac Resynchronization Therapy
  Arms: Cardiac Resynchronization Therapy Group - CRT Group

SUMMARY:
Chagas disease is an endemic problem in Latin America, where millions of people are chronically infected with T. cruzi. Recently, it was assumed to have clinical and epidemiological relevance in several other countries due to migratory and globalizing social factors. CCC occurs in 30-50% of infected individuals, causing considerable morbidity/mortality rates. Heart failure is the most prevalent morbidity. While CRT and drug treatment have been advocated and implemented without much success to improve the clinical condition of patients with CCC, there is no consistent scientific evidence on the role of cardiac contractility modulation (CCM) as a form of adjuvant treatment for heart failure in patients with CCC.

The hypothesis of this study is that patients with CCC, advanced heart failure, severe systolic dysfunction, and non-LBB have better clinical and functional responses when undergoing implantation of a CCM device than when undergoing cardiac resynchronization therapy.

DETAILED DESCRIPTION:
Chagas Disease:

Chagas disease (Trypanosomiasis Americana) is caused by the protozoan parasite Trypanosoma cruzi, which is transmitted to humans through the feces of a hematophagous insect (family Triatominae) in most cases. The infection usually occurs in childhood, and the acute phase has an incubation period of 1 to 2 weeks and can last up to 3 months. Then follows the chronic phase, in which for a long time - 2-4 decades most of the time - patients have only positive serology for Chagas disease (CD), without symptoms or other signs of clinically apparent disease.

Therefore, such patients present the so-called indeterminate form of Chagas disease, whose prognosis is essentially benign.

While due to pathogenic mechanisms still incompletely understood, many patients remain with this form of the disease for life around 30 to 50% of infected individuals evolve to certain forms like cardiac, digestive, or mixed. Chronic Chagas cardiomyopathy (CCC) has a hemodynamic pattern like dilated idiopathic cardiomyopathy but has marked pathophysiological peculiarities. The most common and most serious clinical form of CD is responsible for significant morbidity and mortality in many Latin countries -Americans (and with epidemiological relevance also contemporarily recognized in countries with immigration by individuals from those countries).

It is estimated that 8-10 million people are infected with Trypanosoma cruzi in Latin America and other countries. Considering the worst-case scenario, we can deduce that 3-5 million infected individuals will manifest clinical forms of the disease in its chronic phase.

The disease severity:

In addition to the criteria used in the risk stratification shown in Tables 1 and 2, several markers of worse prognosis have been identified by several authors, especially concerning sudden cardiac death in different clinical contexts.

Characteristics such: as presyncope and syncope; left ventricular dysfunction; heart failure; sustained ventricular tachycardia (VT) or non-sustained ventricular tachycardia; severe bradyarrhythmia (sinus node disease and advanced atrioventricular block); and previous cardiac arrest were identified as markers of risk of sudden cardiac death (SCD). On the other hand, isolated ventricular extrasystoles on Holter monitoring and right bundle-branch block do not significantly interfere with the prognosis of CCC. SCD is often associated with manifestations of heart failure (HF), but it can also occur in patients with asymptomatic left ventricular dysfunction. It accounts for approximately 55 to 65% of all causes of death, whereas refractory HF is a cause of death in about 25 to 30% of patients and systemic or pulmonary thromboembolism in about 10 to 15%. Indicador não definido. Very rarely, aneurysm rupture can be the mechanism of sudden death in CCC.

Recently, the correlation between CCC stages and causes of mortality has been schematically described. SCD usually affects patients from stage II of the disease onwards, being more relevant in stage III and a little less in stage IV, in which refractory heart failure as a cause of death becomes quite frequent.

Therapeutic Options for Heart Failure. As in other heart diseases, the treatment of HF in CCC is based on the routine use of a combination of three types of drugs: diuretics, angiotensin-converting enzyme (ACE) inhibitors, or angiotensin receptor blockers (ARB) and adrenergic beta-blockers (BB). However, despite CD representing an important cause of HF in Latin America, patients with CD and HF were not included in the large studies that validated those drugs to treat HF. Therefore, the real efficacy and tolerability of these drugs in patients with CCC have not been scientifically established, and their use is empirically extrapolated from the support obtained in HF of other etiologies.

In the same sense, the scientific evidence regarding the role of CRT in CCC is not supported by randomized studies. Furthermore, the low prevalence of left bundle block, an independent marker of CRT response, in CCC is a limiting factor for its indication of this therapeutic option. Some observational studies have been carried out to recognize other candidates for CRT in CCC, but the evidence is still poor.

Heart transplantation is a good option for severe cases, but its application is very limited by the low availability of donors.

Recently, an excellent adjunctive option was introduced, and tested in several heart diseases but not in patients with CCC. It is an implantable device capable of modulating myocardial contractility: Cardiac Contractility Modulation (CCM).

Cardiac Contractility Modulation:

CCM consists of high-tension stimulation of the right ventricular septum during the absolute refractory period, 30-40ms after cardiomyocyte activation. This stimulation acts on calcium currents and increases ventricular contractility and, as a consequence, improves functional capacity.

In a 2019 meta-analytic study, Mando R et al. evaluated four randomized studies that applied the CCM technique compared to optimized drug therapy. The authors concluded that, in short-term follow-up, there is health-related quality of life gains (as measured by the Minnesota questionnaire) and that these were significantly greater in patients treated with CCM. However, they did not observe significantly better results in the functional test evaluated by the 6-minute walk test, nor regarding mortality and hospitalization from any causes.

Abraham WT et al. performed an open-label randomized trial to evaluate the adjunctive effect of CCM therapy to optimized therapy in 160 patients with symptoms of HF functional class III or IV by NYHA classification, sinus rhythm, QRS duration <130ms, and LVEF ≥25%, and ≤45%. Of these, 74 patients underwent CCM therapy for 24 weeks. The results indicated that CCM therapy is safe and improves exercise tolerance and quality of life. The composite endpoint of cardiovascular death and HF hospitalizations was also reduced and clinical effects were observed for the entire LVEF range studied. More specifically, superior clinical efficacy was observed in patients with LVEF between 35% and 45%. These data point in the direction that CCM may be an interesting adjuvant option in HF therapy.

Hypothesis:

The hypothesis of this study is that patients with CCC, advanced heart failure, severe systolic dysfunction, and non-LBB have better clinical and functional responses when undergoing implantation of a CCM device than when undergoing cardiac resynchronization therapy.

Objectives:

Primary objective - To assess the short-term impact on quality of life and myocardial contractility of an implantable electronic cardiac device for cardiac contractility modulation compared to CRT in patients with CCC, non-LBBB, and advanced HF.

Secondary objectives - To record the clinical evolution, including the need for hospitalization, the functional class according to the New York Heart Association, and the functional capacity of an implantable electronic cardiac device for cardiac contractility modulation compared to CRT, in patients with CCC, non-LBBB, and advanced HF.

ELIGIBILITY:
Inclusion Criteria:

* Signing of an informed consent form (ICF) before randomization and any study procedure,
* Both genders, age >18 years and <75 years,
* Recent positive (last two years) and documented serology for Chagas disease, in at least two different tests (indirect hemagglutination, indirect immunofluorescence, or ELISA),
* NYHA II-III heart failure functional class,
* LVEF< 35%,
* Non left bundle branch block
* Intraventricular desynchrony (Yu index)
* Global longitudinal strain >11 %.

Exclusion Criteria:

* Participation in another study, presently or terminated <1 year ago, except for a totally unrelated observational study,
* Other concomitant cardiovascular diseases, including uncontrolled diabetes mellitus (systemic arterial hypertension without permitted target organ compromise),
* Kidney dysfunction (serum creatinine >1.5mg/dL or eGFR <30mL/min/1.73m2) or liver dysfunction, with diagnosis of cirrhosis or portal hypertension or elevated serum enzymes (AST or ALT) > 3x the upper limit of normality,
* Moderate or severe chronic obstructive pulmonary disease,
* Peripheral polyneuropathy,
* Hyperthyroidism,
* Current alcoholism or not abandoned for >2 years,
* Diagnosed with psychopathy or psychosis or addiction to illicit drugs,
* Life expectancy <1 year, due to the disease itself or comorbidities (including NYHA class IV),
* Pregnancy or breastfeeding,
* Potential to become pregnant during the study (non-menopausal patients who have not undergone a radical and safe contraceptive process),
* Previously withdrawn from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
QoL Score | At baseline
  KCCQS - Kansas City cardiomyopathy quality score
QoL Score | At 6 months
  KCCQS - Kansas City cardiomyopathy quality score
GLS | At baseline
  Global longitudinal strain at rest/effort - (tissue tracking)
GLS | At 6 months
  Global longitudinal strain at rest/effort - (tissue tracking)

SECONDARY OUTCOMES:
6MWT | At baseline
  6-minute walk test
6MWT | At 6 months
  6-minute walk test
NYHAFC | At baseline
  HF functional class assessed as established by the NYHA
NYHAFC | At 6 months
  HF functional class assessed as established by the NYHA
LVEF | At baseline
  Left ventricle ejection fraction
LVEF | At 6 months
  Left ventricle ejection fraction
Heart Failure Hospitalization (HFH) checklist | Through study completion, an average of 6 months
  Heart Failure Hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- InCor - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dias JC, Kloetzel K. The prognostic value of the electrocardiographic features of chronic Chagas' disease. Rev Inst Med Trop Sao Paulo. 1968 May-Jun;10(3):158-62. No abstract available. PMID 4982469
- [Background] Espinosa R, Carrasco HA, Belandria F, Fuenmayor AM, Molina C, Gonzalez R, Martinez O. Life expectancy analysis in patients with Chagas' disease: prognosis after one decade (1973-1983). Int J Cardiol. 1985 May;8(1):45-56. doi: 10.1016/0167-5273(85)90262-1. PMID 3997291
- [Background] Carrasco HA, Parada H, Guerrero L, Duque M, Duran D, Molina C. Prognostic implications of clinical, electrocardiographic and hemodynamic findings in chronic Chagas' disease. Int J Cardiol. 1994 Jan;43(1):27-38. doi: 10.1016/0167-5273(94)90087-6. PMID 8175216
- [Background] Martinelli Filho M, Sosa E, Nishioka S, Scanavacca M, Bellotti G, Pileggi F. Clinical and electrophysiologic features of syncope in chronic chagasic heart disease. J Cardiovasc Electrophysiol. 1994 Jul;5(7):563-70. doi: 10.1111/j.1540-8167.1994.tb01297.x. PMID 7987526
- [Background] Mady C, Cardoso RH, Barretto AC, da Luz PL, Bellotti G, Pileggi F. Survival and predictors of survival in patients with congestive heart failure due to Chagas' cardiomyopathy. Circulation. 1994 Dec;90(6):3098-102. doi: 10.1161/01.cir.90.6.3098. PMID 7994859
- [Background] Bestetti RB, Dalbo CM, Freitas OC, Teno LA, Castilho OT, Oliveira JS. Noninvasive predictors of mortality for patients with Chagas' heart disease: a multivariate stepwise logistic regression study. Cardiology. 1994;84(4-5):261-7. doi: 10.1159/000176409. PMID 8187110
- [Background] de Paola AA, Gomes JA, Terzian AB, Miyamoto MH, Martinez Fo EE. Ventricular tachycardia during exercise testing as a predictor of sudden death in patients with chronic chagasic cardiomyopathy and ventricular arrhythmias. Br Heart J. 1995 Sep;74(3):293-5. doi: 10.1136/hrt.74.3.293. PMID 7547025
- [Background] Bestetti RB, Dalbo CM, Arruda CA, Correia Filho D, Freitas OC. Predictors of sudden cardiac death for patients with Chagas' disease: a hospital-derived cohort study. Cardiology. 1996 Nov-Dec;87(6):481-7. doi: 10.1159/000177142. PMID 8904674
- [Background] Carrasco HA, Guerrero L, Parada H, Molina C, Vegas E, Chuecos R. Ventricular arrhythmias and left ventricular myocardial function in chronic chagasic patients. Int J Cardiol. 1990 Jul;28(1):35-41. doi: 10.1016/0167-5273(90)90006-q. PMID 2365530
- [Background] Lopes ER. Sudden death in patients with Chagas disease. Mem Inst Oswaldo Cruz. 1999;94 Suppl 1:321-4. doi: 10.1590/s0074-02761999000700061. No abstract available. PMID 10677747
- [Background] Rassi A Jr, Rassi SG, Rassi A. Sudden death in Chagas' disease. Arq Bras Cardiol. 2001 Jan;76(1):75-96. doi: 10.1590/s0066-782x2001000100008. No abstract available. English, Portuguese. PMID 11175486
- [Background] Bestetti R. Stroke in a hospital-derived cohort of patients with chronic Chagas' disease. Acta Cardiol. 2000 Feb;55(1):33-8. doi: 10.2143/AC.55.1.2005715. PMID 10707756
- [Background] Carod-Artal FJ, Vargas AP, Horan TA, Nunes LG. Chagasic cardiomyopathy is independently associated with ischemic stroke in Chagas disease. Stroke. 2005 May;36(5):965-70. doi: 10.1161/01.STR.0000163104.92943.50. Epub 2005 Apr 21. PMID 15845889
- [Background] Sousa AS, Xavier SS, Freitas GR, Hasslocher-Moreno A. Prevention strategies of cardioembolic ischemic stroke in Chagas' disease. Arq Bras Cardiol. 2008 Nov;91(5):306-10. doi: 10.1590/s0066-782x2008001700004. English, Portuguese. PMID 19142374
- [Background] Oliveira JS, Barbieri Neto J. [Chagasic cardiopathy. Rupture of the apical aneurysm]. Arq Bras Cardiol. 1970 Oct;23(5):335-8. No abstract available. Portuguese. PMID 4994717
- [Background] Pinto Dias JC. [Natural history of Chagas disease]. Arq Bras Cardiol. 1995 Oct;65(4):359-66. No abstract available. Portuguese. PMID 8728813
- [Background] Rassi A Jr, Rassi A, Marin-Neto JA. Chagas disease. Lancet. 2010 Apr 17;375(9723):1388-402. doi: 10.1016/S0140-6736(10)60061-X. PMID 20399979
- [Background] Dias JC. The indeterminate form of human chronic Chagas' disease A clinical epidemiological review. Rev Soc Bras Med Trop. 1989 Jul-Sep;22(3):147-56. doi: 10.1590/s0037-86821989000300007. PMID 2486527
- [Background] Barretto AC, Ianni BM. The undetermined form of Chagas' heart disease: concept and forensic implications. Sao Paulo Med J. 1995 Mar-Apr;113(2):797-801. doi: 10.1590/s1516-31801995000200010. PMID 8650479
- [Background] Marin-Neto JA, Cunha-Neto E, Maciel BC, Simoes MV. Pathogenesis of chronic Chagas heart disease. Circulation. 2007 Mar 6;115(9):1109-23. doi: 10.1161/CIRCULATIONAHA.106.624296. PMID 17339569
- [Background] Schmunis GA. Epidemiology of Chagas disease in non-endemic countries: the role of international migration. Mem Inst Oswaldo Cruz. 2007 Oct 30;102 Suppl 1:75-85. doi: 10.1590/s0074-02762007005000093. PMID 17891282
- [Background] Dias JC, Prata A, Correia D. Problems and perspectives for Chagas disease control: in search of a realistic analysis. Rev Soc Bras Med Trop. 2008 Mar-Apr;41(2):193-6. doi: 10.1590/s0037-86822008000200012. PMID 18545843
- [Background] Moncayo A, Silveira AC. Current epidemiological trends for Chagas disease in Latin America and future challenges in epidemiology, surveillance and health policy. Mem Inst Oswaldo Cruz. 2009 Jul;104 Suppl 1:17-30. doi: 10.1590/s0074-02762009000900005. PMID 19753454
- [Background] Rassi A Jr, Dias JC, Marin-Neto JA, Rassi A. Challenges and opportunities for primary, secondary, and tertiary prevention of Chagas' disease. Heart. 2009 Apr;95(7):524-34. doi: 10.1136/hrt.2008.159624. Epub 2009 Jan 8. PMID 19131444
- [Background] Rassi A Jr, Rassi A, Little WC, Xavier SS, Rassi SG, Rassi AG, Rassi GG, Hasslocher-Moreno A, Sousa AS, Scanavacca MI. Development and validation of a risk score for predicting death in Chagas' heart disease. N Engl J Med. 2006 Aug 24;355(8):799-808. doi: 10.1056/NEJMoa053241. PMID 16928995
- [Background] Brunckhorst CB, Shemer I, Mika Y, Ben-Haim SA, Burkhoff D. Cardiac contractility modulation by non-excitatory currents: studies in isolated cardiac muscle. Eur J Heart Fail. 2006 Jan;8(1):7-15. doi: 10.1016/j.ejheart.2005.05.011. Epub 2005 Oct 3. PMID 16202650
- [Background] Kahwash R, Burkhoff D, Abraham WT. Cardiac contractility modulation in patients with advanced heart failure. Expert Rev Cardiovasc Ther. 2013 May;11(5):635-45. doi: 10.1586/erc.13.48. PMID 23621145
- [Background] Abi-Samra F, Gutterman D. Cardiac contractility modulation: a novel approach for the treatment of heart failure. Heart Fail Rev. 2016 Nov;21(6):645-660. doi: 10.1007/s10741-016-9571-6. PMID 27394714
- [Background] Mando R, Goel A, Habash F, Saad M, Ayoub K, Vallurupalli S, Maskoun W. Outcomes of Cardiac Contractility Modulation: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Cardiovasc Ther. 2019 Jun 17;2019:9769724. doi: 10.1155/2019/9769724. eCollection 2019. PMID 31772622
- [Background] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- [Background] Hinkle LE Jr, Thaler HT. Clinical classification of cardiac deaths. Circulation. 1982 Mar;65(3):457-64. doi: 10.1161/01.cir.65.3.457. PMID 7055867
- [Background] Parissis JT, Nikolaou M, Farmakis D, Paraskevaidis IA, Bistola V, Venetsanou K, Katsaras D, Filippatos G, Kremastinos DT. Self-assessment of health status is associated with inflammatory activation and predicts long-term outcomes in chronic heart failure. Eur J Heart Fail. 2009 Feb;11(2):163-9. doi: 10.1093/eurjhf/hfn032. PMID 19168514